CLINICAL TRIAL: NCT01309854
Title: An Open-Label, Single Center Study to Assess the Pharmacokinetics of Pioglitazone in Healthy Subjects When Administered Alone and in Combination With Fostamatinib 100 mg Twice Daily
Brief Title: Effects of Administration of Fostamatinib on Blood Concentrations of Pioglitazone in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Layton / Medical Science Director, AstraZeneca
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00014
Record Dates: First submitted 2011-02-21; First posted 2011-03-07 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Rheumatoid Arthritis; Healthy Volunteers; Pharmacokinetics; Pioglitazone; Drug-drug Interaction; Amount of Pioglitazone in Blood
Keywords: Phase 1; healthy volunteers; pharmacokinetics; Rheumatoid arthritis; RA; fostamatinib; pioglitazone; drug-drug interaction
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib; Pioglitazone

ARMS (2):
- pioglitazone (Experimental)
  Interventions: Drug: fostamatinib; Drug: pioglitazone
- pioglitazone and fostamatinib (Experimental)
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: fostamatinib — oral tablets, 100mg (2 X 50mg) twice daily for 8 days
  Arms: pioglitazone
Drug: pioglitazone — oral tablets, 30mg single dose per period

SUMMARY:
The purpose of this study is to investigate the drug interaction between fostamatinib and pioglitazone by comparing the safety, tolerability and plasma concentration of pioglitazone when administered alone and with fostamatinib in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Males or females (of non-child bearing potential) aged 18 to 55 years (inclusive)
* Minimum weight of 50 kg and a body mass index (BMI) of 18 to 35 kg/m2 (inclusive)
* Males must be willing to use barrier contraception ie, condoms, from the first administration until 2 weeks after the last administration of the investigational product

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic or renal disease (except for cholecystectomy)
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of the investigational product
* Subjects who smoke more than 5 cigarettes or the equivalent in tobacco per day
* Absolute neutrophil count of less than 2500/mm3 or 2.5 x 109/L
* Any previous treatment with fostamatinib or pioglitazone

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To assess pharmacokinetics (PK) of pioglitazone including but not limited to AUC and Cmax | Period 1: Pre-dose to 48h post dose
To assess pharmacokinetics (PK) of pioglitazone including but not limited to AUC and Cmax | Period 2: Pre-dose to 48h post dose

SECONDARY OUTCOMES:
To assess pharmacokinetics (PK) of hydroxypioglitazone (active metabolite) including but not limited to AUC and Cmax | Period 1: Pre-dose to 48h post dose
To assess pharmacokinetics (PK) of hydroxypioglitazone (active metabolite) including but not limited to AUC and Cmax | Period 2: Pre-dose to 48h post dose
To examine the safety and tolerability | From screening, Day -1 to Day 9 and follow up visit (Day 16)
  To examine the safety and tolerability of fostamatinib in combination with pioglitazone. Assessments include: Adverse events, laboratory assessments, vital signs, physical examination and 12-lead electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, MD, MRCP, Study Director — AstraZeneca; Carlos Prendes, MD, Principal Investigator — Quintiles Overland Park, Phase 1 Unit
Locations (1):
- Research Site, Overland Park, Kansas, United States